CLINICAL TRIAL: NCT02194140
Title: Improvement of Appendix Identification and Appendicitis Diagnosis in Ultrasound After Administration of Iodinated Oral Contrast Medium
Brief Title: Improvement of Appendix Identification and Appendicitis Diagnosis in us After Administration of Oral Contrast Medium
Acronym: us
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 028-14
Record Dates: First submitted 2014-06-28; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Appendicitis
Keywords: ultrasound; iodinated contrast material; computed tomography
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oral contrast (Other): oral iodinated contrast material
  Interventions: Other: oral iodinated contrast material

INTERVENTIONS:
Other: oral iodinated contrast material — diluted in water
  Other Names: telebrix 35

SUMMARY:
Rate of appendix localization on ultrasound is not high. We suggest a way to improve it's localization by oral administration of iodinated contrast material.

DETAILED DESCRIPTION:
The administration of oral iodinated contrast material might facilitate identification of the appendix and accurate diagnosis of appendicitis. When indicated will shorten time to CT examination.

ELIGIBILITY:
Inclusion Criteria:

* patients in emergency department with right lower quadrant pain

Exclusion Criteria:

* patients under 18 years old
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Appendix identification rate on ultrasound | At the time of ultrasound examination up to 1 hour
  Positive identification of the appendix by ultrasound croteria

SECONDARY OUTCOMES:
improved rate of correctly diagnosed appendicitis | At time of surgery or patholoy results if available within 14 days
  Results acording to surgery or patholoy reports

OTHER OUTCOMES:
shortening waiting time for CT | At time of CT examination up to 1 hour
  Measuring time from referal to examination

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Reindorp, MD, Principal Investigator — Hillel Yaffe Medical Center Hadera Israel
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Background] Trout AT, Sanchez R, Ladino-Torres MF, Pai DR, Strouse PJ. A critical evaluation of US for the diagnosis of pediatric acute appendicitis in a real-life setting: how can we improve the diagnostic value of sonography? Pediatr Radiol. 2012 Jul;42(7):813-23. doi: 10.1007/s00247-012-2358-6. Epub 2012 Mar 9. PMID 22402833